CLINICAL TRIAL: NCT05672667
Title: A Pharmacokinetic Study of Intravenous and Intranasal Oxytocin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00089938; 1P01NS119159-01A1 (NIH)
Record Dates: First submitted 2022-12-20; First posted 2023-01-05 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2023-12

CONDITIONS: Healthy Volunteer Study
Keywords: Acute Pain; Chronic Pain; Intravenous Oxytocin; Intranasal Oxytocin
MeSH Terms: conditions — Acute Pain; Chronic Pain | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Each subject will receive 14 micrograms of oxytocin intravenously over 30 minutes and 102 micrograms of oxytocin intranasally.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oxytocin Administration (Intravenous, then Intranasal) (Experimental): Oxytocin 14 micrograms infusion over 30 minutes on first study day. Oxytocin 102 micrograms by intranasal spray on second study day.
  Interventions: Drug: intravenous oxytocin; Drug: intranasal oxytocin

INTERVENTIONS:
Drug: intravenous oxytocin — Oxytocin given by intravenous route
  Other Names: Pitocin
Drug: intranasal oxytocin — Oxytocin given by intranasal administration
  Other Names: TNX-1900

SUMMARY:
The main purpose of this study is to sample blood and model the plasma pharmacokinetics (PK) of a single dose of intravenous (IV) oxytocin and a single dose of intranasal (i.n.) oxytocin.

This is an unblinded study of subjects, all of whom will receive an intravenous (IV) infusion and intranasal (i.n.) dose of oxytocin (a naturally occurring hormone that is made in the brain) with blood samples taken thereafter in order to create a formula to describe the concentrations of oxytocin in the blood over time (pharmacokinetics).

In this study healthy volunteers and people are recruited for a two day study. Each study participant will have 2 IV catheters placed (one in each arm) for the day of IV oxytocin dosing and 1 IV catheter on the day of i.n. oxytocin dosing. After placement of the IV catheters, an infusion of oxytocin will be given over a 30 minute period. Blood samples will be taken after the infusion begins and several times during and after the infusion. The blood will be drawn through the IV catheter not used for the oxytocin infusion. For the intranasal oxytocin administration day, 1 IV catheter will be placed and several blood samples will be taken after administration.

DETAILED DESCRIPTION:
This is an unblinded, sequential study of subjects; all participants will receive an infusion of oxytocin and intranasal administration of oxytocin with blood samples taken thereafter in order to create a formula to describe the concentrations of oxytocin in the blood over time (pharmacokinetics). In this study healthy volunteers. Participants will come to the Clinical Research Unit (CRU) on study day 1 and have two IVs inserted; one in each arm. Participants will get a 30 minute infusion through one of the IV catheters of oxytocin and blood will be taken several times over the next 120 minutes, plasma separated, and the amount of oxytocin measured in the plasma samples. Participants will come to the CRU on study day 2 and have one IV inserted; in the arm. Participants will self administer intranasal oxytocin and blood will be taken several times over the next 60 minutes and the amount of oxytocin measured in the plasma samples. This information will be analyzed by another group at Stanford University under a data sharing agreement between the institutions and funded by a grant from the National Institutes of Health. Compartmental modeling will be performed using NONMEM to describe the change in oxytocin concentrations over time. The effect of subject age, sex, race, ethnicity and weight on the pharmacokinetics of oxytocin will be examined, since these factors can affect pharmacokinetics and are important to better adjust the dose of drug to the individual.

The main purpose of this study is to determine the amount of oxytocin in plasma after IV and i.n. administration.

The research participants will not benefit from this study, but the knowledge investigators get will be important to adjust oxytocin dose to individuals, and to be able to calculate plasma oxytocin concentrations after various doses in the future. The sample size chosen is needed to get an accurate estimate for the parameters in the pharmacokinetic model for the population, not just the subjects in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female > 18 and < 75 years of age, Body Mass Index (BMI) <40.
* Generally in good health as determined by the Principal Investigator based on prior medical history, American Society of Anesthesiologists physical status 1 or 2.
* For healthy volunteers, normal blood pressure (systolic 100-140 mmHg; diastolic 60-90 mmHg) resting heart rate 45-90 beats per minute) without medication. For those with hypertension, blood pressure controlled with anti-hypertensive medication and with a resting heart rate 45-100 beats per minute.
* Female subjects of child-bearing potential and those < 1 year post-menopausal, must be practicing highly effective methods of birth control such as hormonal methods (e.g., combined oral, implantable, injectable, or transdermal contraceptives), double barrier methods (e.g., condoms, sponge, diaphragm, or vaginal ring plus spermicidal jellies or cream), or total abstinence from heterosexual intercourse for a minimum of 1 full cycle before study drug administration.

Exclusion Criteria:

* Hypersensitivity, allergy, or significant reaction to any ingredient of Pitocin®
* Any disease, diagnosis, or condition (medical or surgical) that, in the opinion of the Principal Investigator, would place the subject at increased risk (active gynecologic disease in which increased tone would be detrimental e.g., uterine fibroids with ongoing bleeding), compromise the subject's compliance with study procedures, or compromise the quality of the data
* Women who are pregnant (positive result for urine pregnancy test at visit 1), women who are currently nursing or lactating, women that have been pregnant within 2 years
* Subjects with neuropathy, chronic pain (being treated on a daily basis), diabetes mellitus, or taking benzodiazepines or pain medications on a daily basis.
* Subjects with current or history of ventricular tachycardia, atrial fibrillation or prolonged QT interval.
* Subjects with past or current history of hyponatremia or at risk for hyponatremia; anyone taking thiazide diuretics, loop diuretics, combination diuretics, lithium, carbamazepine, enalapril, Ramipril, celecoxib, temazepam, gliclazide, glimepiride, glibenclamide, glipizide, omeprazole, pantoprazole, desmopressin, Selective serotonin reuptake inhibitors (SSRI's) , Monoamine oxidase inhibitors (MAOI), or the recreational drug ecstasy.
* Subjects with a known latex allergy.
* History of chronic nasal obstruction or local pathology in nostril pathway which, in the opinion of the investigator, would prevent appropriate nasal administration of the study drug.
* Use of over the counter nasal products (ie. Saline spray, Neti-Pot, etc.) or intranasal corticosteroid medications during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C Eisenach, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan Description: Statistical programs in the data analysis will be written in R. The software and anonymized data will be included both as digital supplements in the published papers and will be posted on GitHub under github.com/StevenLShafer. Interested investigators will be able to reproduce the published analyses from these files. Consistent with the posting of software and data to the OpenTCI initiative, the software and de-identified data will be made available with "no strings attached," enabling investigators to freely use the data to inform or supplement additional research without restriction. Data to be made available are oxytocin dose, times of sampling (relative to the start of dosing), plasma oxytocin concentrations at those times for each subject, and age, weight, and sex for each subject.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will become available upon publication or upon posting results in ClinicalTrials.gov, whichever comes first, with no expiration.
Access Criteria: These data are freely shared to all and will be posted at the URL below
URL: https://github.com/StevenLShafer

REFERENCES:
- [Derived] Shafer SL, Ririe DG, Miller S, Curry RS, Hsu DT, Sullivan GM, Eisenach JC. Plasma pharmacokinetics of intravenous and intranasal oxytocin in nonpregnant adults. Br J Anaesth. 2025 May;134(5):1513-1522. doi: 10.1016/j.bja.2024.12.046. Epub 2025 Mar 21. PMID 40121179

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled between February, 2023 and August, 2023, and were recruited by IRB approved advertisements in the local community as well as direct contacting in a list of subjects who requested they be contacted regarding new research studies.
Period: Overall Study
Arm/Group | Oxytocin Administration (Intravenous, Then Intranasal)
Started | 25
Completed | 24
Not Completed | 1
Not completed — Vasovagal reaction with IV cannulation. Oxytocin was not infused and subject was withdrawn. | 1

BASELINE CHARACTERISTICS:
Population: 25 subjects consented to participate and provided baseline data, but one individual was withdrawn after a vasovagal event on insertion of IV cannula and did not receive oxytocin IV or intranasally.
Arm/Group | Oxytocin Administration (Intravenous, Then Intranasal)
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Plasma Oxytocin Concentration 2 Minutes After Infusion Initiated
Description: Blood will be sampled at specified intervals during and after the infusion. Plasma will be separated, rapidly frozen, and later analyzed for oxytocin concentration
Time Frame: 2 minutes after oxytocin infusion initiated
Measure: Mean (Standard Deviation); unit: picograms/ml of oxytocin
Arm/Group | Oxytocin Administration (Intravenous, Then Intranasal)
Number analyzed (Participants) | 24
picograms/ml of oxytocin | 105 (47)

2. Primary Outcome: Plasma Oxytocin Concentration 5 Minutes After Infusion Initiated
Description: as for outcome 1
Time Frame: 5 minutes after oxytocin infusion initiated
Measure: Mean (Standard Deviation); unit: picograms/ml of oxytocin
Arm/Group | Oxytocin Administration (Intravenous, Then Intranasal)
Number analyzed (Participants) | 24
picograms/ml of oxytocin | 257 (80)

3. Primary Outcome: Plasma Oxytocin Concentration 10 Minutes After Infusion Initiated
Description: as for outcome 1
Time Frame: 10 minutes after oxytocin infusion initiated
Measure: Mean (Standard Deviation); unit: picograms/ml of oxytocin
Arm/Group | Oxytocin Administration (Intravenous, Then Intranasal)
Number analyzed (Participants) | 24
picograms/ml of oxytocin | 365 (77)

4. Primary Outcome: Plasma Oxytocin Concentration 20 Minutes After Infusion Initiated
Description: as for outcome 1
Time Frame: 20 minutes after oxytocin infusion initiated
Measure: Mean (Standard Deviation); unit: picograms/ml of oxytocin
Arm/Group | Oxytocin Administration (Intravenous, Then Intranasal)
Number analyzed (Participants) | 24
picograms/ml of oxytocin | 452 (89)

5. Primary Outcome: Plasma Oxytocin Concentration 30 Minutes After Infusion Initiated
Description: as for outcome 1
Time Frame: 30 minutes after oxytocin infusion initiated
Measure: Mean (Standard Deviation); unit: picograms/ml of oxytocin
Arm/Group | Oxytocin Administration (Intravenous, Then Intranasal)
Number analyzed (Participants) | 24
picograms/ml of oxytocin | 462 (139)

6. Primary Outcome: Plasma Oxytocin Concentration 40 Minutes After Infusion Initiated
Description: as for outcome 1
Time Frame: 40 minutes after oxytocin infusion initiated
Measure: Mean (Standard Deviation); unit: picograms/ml of oxytocin
Arm/Group | Oxytocin Administration (Intravenous, Then Intranasal)
Number analyzed (Participants) | 24
picograms/ml of oxytocin | 193 (79)

7. Primary Outcome: Plasma Oxytocin Concentration 50 Minutes After Infusion Initiated
Description: as for outcome 1
Time Frame: 50 minutes after oxytocin infusion initiated
Measure: Mean (Standard Deviation); unit: picograms/ml of oxytocin
Arm/Group | Oxytocin Administration (Intravenous, Then Intranasal)
Number analyzed (Participants) | 24
picograms/ml of oxytocin | 118 (73)

8. Primary Outcome: Plasma Oxytocin Concentration 65 Minutes After Infusion Initiated
Description: as for outcome 1
Time Frame: 65 minutes after oxytocin infusion initiated
Measure: Mean (Standard Deviation); unit: picograms/ml of oxytocin
Arm/Group | Oxytocin Administration (Intravenous, Then Intranasal)
Number analyzed (Participants) | 24
picograms/ml of oxytocin | 51 (21)

9. Primary Outcome: Plasma Oxytocin Concentration 90 Minutes After Infusion Initiated
Description: as for outcome 1
Time Frame: 90 minutes after oxytocin infusion initiated
Measure: Mean (Standard Deviation); unit: picograms/ml of oxytocin
Arm/Group | Oxytocin Administration (Intravenous, Then Intranasal)
Number analyzed (Participants) | 24
picograms/ml of oxytocin | 23 (10)

10. Primary Outcome: Plasma Oxytocin Concentration 120 Minutes After Infusion Initiated
Description: as for outcome 1
Time Frame: 120 minutes after oxytocin infusion initiated
Measure: Mean (Standard Deviation); unit: picograms/ml of oxytocin
Arm/Group | Oxytocin Administration (Intravenous, Then Intranasal)
Number analyzed (Participants) | 24
picograms/ml of oxytocin | 11 (6)

11. Primary Outcome: Plasma Oxytocin Concentration 1 Minute After First Intranasal Puffs
Description: Blood will be sampled at specified intervals after the intranasal administration of oxytocin. Plasma will be separated, rapidly frozen, and later analyzed for oxytocin concentration
Time Frame: 1 minute after intranasal oxytocin administration
Population: Samples were obtained from 24 subjects, but only 9 had oxytocin concentrations above the limit of detection of the assay (2 pg/mL).
Measure: Mean (Standard Deviation); unit: picograms/ml of oxytocin
Arm/Group | Oxytocin Administration (Intravenous, Then Intranasal)
Number analyzed (Participants) | 9
picograms/ml of oxytocin | 3.4 (1.1)

12. Primary Outcome: Plasma Oxytocin Concentration 2 Minutes After First Intranasal Puffs
Description: as for outcome 11
Time Frame: 2 minutes after intranasal oxytocin administration
Population: Samples were obtained from 24 subjects, but only 14 had oxytocin concentrations above the limit of detection of the assay (2 pg/mL).
Measure: Mean (Standard Deviation); unit: picograms/ml of oxytocin
Arm/Group | Oxytocin Administration (Intravenous, Then Intranasal)
Number analyzed (Participants) | 14
picograms/ml of oxytocin | 11.7 (6.6)

13. Primary Outcome: Plasma Oxytocin Concentration 5 Minutes After First Intranasal Puffs
Description: as for outcome 11
Time Frame: 5 minutes after intranasal oxytocin administration
Measure: Mean (Standard Deviation); unit: picograms/ml of oxytocin
Arm/Group | Oxytocin Administration (Intravenous, Then Intranasal)
Number analyzed (Participants) | 24
picograms/ml of oxytocin | 14.2 (11.5)

14. Primary Outcome: Plasma Oxytocin Concentration 7 Minutes After First Intranasal Puffs
Description: as for outcome 11
Time Frame: 7 minutes after intranasal oxytocin administration
Measure: Mean (Standard Deviation); unit: picograms/ml of oxytocin
Arm/Group | Oxytocin Administration (Intravenous, Then Intranasal)
Number analyzed (Participants) | 24
picograms/ml of oxytocin | 23.5 (15.7)

15. Primary Outcome: Plasma Oxytocin Concentration 10 Minutes After First Intranasal Puffs
Description: as for outcome 11
Time Frame: 10 minutes after intranasal oxytocin administration
Measure: Mean (Standard Deviation); unit: picograms/ml of oxytocin
Arm/Group | Oxytocin Administration (Intravenous, Then Intranasal)
Number analyzed (Participants) | 24
picograms/ml of oxytocin | 26.5 (15.3)

16. Primary Outcome: Plasma Oxytocin Concentration 15 Minutes After First Intranasal Puffs
Description: as for outcome 11
Time Frame: 15 minutes after intranasal oxytocin administration
Measure: Mean (Standard Deviation); unit: picograms/ml of oxytocin
Arm/Group | Oxytocin Administration (Intravenous, Then Intranasal)
Number analyzed (Participants) | 24
picograms/ml of oxytocin | 24.5 (17.5)

17. Primary Outcome: Plasma Oxytocin Concentration 20 Minutes After First Intranasal Puffs
Description: as for outcome 11
Time Frame: 20 minutes after intranasal oxytocin administration
Measure: Mean (Standard Deviation); unit: picograms/ml of oxytocin
Arm/Group | Oxytocin Administration (Intravenous, Then Intranasal)
Number analyzed (Participants) | 24
picograms/ml of oxytocin | 21 (15.5)

18. Primary Outcome: Plasma Oxytocin Concentration 25 Minutes After First Intranasal Puffs
Description: as for outcome 11
Time Frame: 25 minutes after intranasal oxytocin administration
Measure: Mean (Standard Deviation); unit: picograms/ml of oxytocin
Arm/Group | Oxytocin Administration (Intravenous, Then Intranasal)
Number analyzed (Participants) | 24
picograms/ml of oxytocin | 18.6 (14.8)

19. Primary Outcome: Plasma Oxytocin Concentration 35 Minutes After First Intranasal Puffs
Description: as for outcome 11
Time Frame: 35 minutes after intranasal oxytocin administration
Population: Samples were obtained from 24 subjects, but only 23 had oxytocin concentrations above the limit of detection of the assay (2 pg/mL).
Measure: Mean (Standard Deviation); unit: picograms/ml of oxytocin
Arm/Group | Oxytocin Administration (Intravenous, Then Intranasal)
Number analyzed (Participants) | 23
picograms/ml of oxytocin | 20.1 (32.4)

20. Primary Outcome: Plasma Oxytocin Concentration 45 Minutes After First Intranasal Puffs
Description: as for outcome 11
Time Frame: 45 minutes after intranasal oxytocin administration
Population: Samples were obtained from 24 subjects, but only 22 had oxytocin concentrations above the limit of detection of the assay (2 pg/mL).
Measure: Mean (Standard Deviation); unit: picograms/ml of oxytocin
Arm/Group | Oxytocin Administration (Intravenous, Then Intranasal)
Number analyzed (Participants) | 22
picograms/ml of oxytocin | 10.8 (8.0)

21. Primary Outcome: Plasma Oxytocin Concentration 60 Minutes After First Intranasal Puffs
Description: as for outcome 11
Time Frame: 60 minutes after intranasal oxytocin administration
Population: Samples were obtained from 24 subjects, but only 21 had oxytocin concentrations above the limit of detection of the assay (2 pg/mL).
Measure: Mean (Standard Deviation); unit: picograms/ml of oxytocin
Arm/Group | Oxytocin Administration (Intravenous, Then Intranasal)
Number analyzed (Participants) | 21
picograms/ml of oxytocin | 7.2 (5.1)

ADVERSE EVENTS:
Time Frame: 1 week after intravenous oxytocin and 1 week after intranasal oxytocin.
Groups:
- Intravenous Oxytocin Infusion Study Day: Oxytocin 14 micrograms infusion over 30 minutes on first study day.
- Intranasal Oxytocin Spray Study Day: Oxytocin 102 micrograms by intranasal spray on second study day.
Arm/Group | Intravenous Oxytocin Infusion Study Day | Intranasal Oxytocin Spray Study Day
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 4/24 | 3/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Oxytocin Infusion Study Day (N=24) | Intranasal Oxytocin Spray Study Day (N=24)
Feeling of warmth after intravenous oxytocin (General disorders) | 3 (3) | 0 (0) — Feeling of warmth which was neither painful nor unpleasant, beginning 2 min after start of oxytocin infusion, lasting 2 minutes
Red face after intravenous oxytocin (Vascular disorders) | 1 (1) | 0 (0) — Facial redness and flushing which was neither painful nor unpleasant, beginning 1 min after starting oxytocin infusion, lasting 1 min.
Rhinorrhea after intranasal oxytocin (General disorders) | 0 (0) | 2 (2) — Clear rhinorrhea lasting 4 min in one case and 6 hr in another after intranasal oxytocin
Sternutation after intranasal oxytocin (General disorders) | 0 (0) | 2 (2) — Single sneeze occuring one min after intranasal spray

LIMITATIONS AND CAVEATS:
Generalizability is limited by the single center design, lack of severely obese subjects, and, despite recruitment efforts, lack of race and ethnic diversity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-27): https://cdn.clinicaltrials.gov/large-docs/67/NCT05672667/Prot_SAP_001.pdf
  • Informed Consent Form (2023-02-06): https://cdn.clinicaltrials.gov/large-docs/67/NCT05672667/ICF_000.pdf